CLINICAL TRIAL: NCT00005881
Title: Assessment of Health/Quality of Life in Survivors of Childhood Cancer
Brief Title: Quality of Life in Children Treated for Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AS972; CCG-AS972 (Other: Children's Cancer Group); CCG-S9702 (Other: Children's Cancer Group); NCI-P00-0148 (Other: NCI Trial Identifier); CDR0000067920 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-06-02; First posted 2004-02-02 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood acute lymphoblastic leukemia; childhood Burkitt lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; unspecified childhood solid tumor, protocol specific; childhood acute myeloid leukemia in remission; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of life forms: Completion of the development of an instrument [Minneapolis-Manchester Quality of Life (MM-QOL)] that measures HRQOL in the survivors of childhood cancer in a standardized, valid way and to assess the feasibility of incorporating this endpoint in a variety of clinical trials.
  Interventions: Other: Quality of Life Forms

INTERVENTIONS:
Other: Quality of Life Forms — Completion of the instrument [Minneapolis-Manchester Quality of Life (MM-QOL)] that measures HRQOL in the survivors of childhood cancer in a standardized, valid way and to assess the feasibility of incorporating this endpoint in a variety of clinical trials.

SUMMARY:
RATIONALE: Questionnaires that measure quality of life may improve the ability to plan treatment for children with cancer.

PURPOSE: This randomized clinical trial is studying the quality of life in children treated for cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the validity and reliability of a quality of life questionnaire (MM-QOL) that is being developed for patients with previously or currently treated childhood cancers.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (8-12 vs 13-20) and treatment (current vs previous). Patients are randomized to one of two arms of the study. Arm I (Reliability): Patients will complete the same questionnaire two weeks apart. (age 13-20 stratum closed as of 7/14/00) Arm II (Validity): Patients will complete a study questionnaire plus a Child Health Questionnaire. Patients between ages 8-12 are interviewed and patients between ages 13-20 complete a written questionnaire.

PROJECTED ACCRUAL: A total of 716 patients (416 for arm I (208 for 8-12 age group and 208 for 13-20 age group) and 300 for arm II (150 for 8-12 age group and 150 for 13-20 age group)) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Prior or current diagnosis of any pediatric cancer Current chemoradiotherapy (at least 2 months since start of therapy) OR At least 1 year since prior treatment and in remission

PATIENT CHARACTERISTICS: Age: 8 to 20 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Previous treatment for cancer or currently undergoing treatment for cancer.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2000-04; Primary Completion 2003-03 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | Length of study
  To complete the development of a self-reported, quality of life questionnaire (MM-QOL) for the pediatric oncology population.

SECONDARY OUTCOMES:
To see if this measure will discriminate between i) those undergoing treatment for cancer, ii) those who are survivors of cancer, and iii) a national sample of age- and sex-matched controls. | Length of study
  To assess the validity of a quality of life questionnaire (MM-QOL) that is being developed for survivors of childhood cancer. To see if this measure will discriminate between i) those undergoing treatment for cancer, ii) those who are survivors of cancer, and iii) a national sample of age- and sex-matched controls (data has already been collected on the latter). To compare the responses to the new scale items with those from established scales (CHQ) that tap relevant QOL domains such as emotional, social, and physical functioning.
Test internal scale reliability | Length of study
  To assess the reliability of a quality of life questionnaire (MM-QOL) that is being developed for the survivors of childhood cancer. To test internal scale reliability (studies already being conducted). To assess test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, MD, MPH, Study Chair — City of Hope Comprehensive Cancer Center
Locations (17):
- United States (17):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin